CLINICAL TRIAL: NCT02934646
Title: Clinical Validation of a Powered Exoskeleton for the Treatment of Elbow Spasticity: Phase II Study
Brief Title: Powered Exoskeleton for the Treatment of Elbow Spasticity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auxilium Vitae Volterra (Other)
Collaborators: Azienda USL Toscana Nord Ovest (Other); Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN20161
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Muscle Spasticity; Stroke
Keywords: Robotics; Upper Extremity
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subacute stroke patients (Experimental): Elbow passive/active robotic treatment provided by NEUROExos Elbow Module
  Interventions: Device: Robotic treatment

INTERVENTIONS:
Device: Robotic treatment — Passive/active elbow mobilizzation provided by NEUROExos Elbow Module Robotic device

SUMMARY:
This is a phase-II clinical study to assess whether intense passive mobilization of the elbow during the early stage is effective in preventing spasticity from occurring at a later stage. A group of subacute stroke patients was treated with the device named NEUROExos Elbow Module (NEEM) on a daily basis, in addition to traditional physical therapy. The outcome was assessed in terms of (i) system safety, (ii) system usability and (iii) treatment efficacy.

Investigators expected that intense therapy performed in the sub-acute phase following the stroke would be effective in preventing elbow spasticity from occurring at a later stage (i.e. 3-4 months after the stroke), the latter being quantified by means of the Modified Ashworth Scale (MAS). Similarly to other phase-II studies in the field of post-stroke rehabilitation, the present study will include only one group of patients. As a secondary objective, similarly to other studies with robot-assisted therapy, investigators wiil test the ability of this system to be used for assessing rehabilitation outcome. Investigators will introduce novel evaluation metrics based on the kinematics and kinetics variables recorded by the NEEM and compared them with MAS values.

ELIGIBILITY:
Inclusion Criteria:

1. Upper limb spasticity due to neurological impairment;
2. Cognitive abilities sufficient for understanding instructions;
3. Absence of severe pain assessed as Visual Analogic Score (VAS) < 4 (range 0-10).

Exclusion Criteria:

1. Unstable general clinical conditions;
2. Unability to keep sitting posture;
3. Tendon retractions limiting upper limb joints range of motion.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 2 weeks
  Impairmente level maesure according to ICF

SECONDARY OUTCOMES:
Range of Motion | 2 weeks
  Impairmente level maesure according to ICF
Maximum Extension Torque | 2 weeks
  Paramenter directly exterted by the device
Zero-Torque Angle | 2 weeks
  Paramenter directly exterted by the device

IPD SHARING:
Plan to Share IPD: No